CLINICAL TRIAL: NCT03090958
Title: AllyQuest: Engaging HIV+ YMSM in Care Through Social Networking and Gamification
Acronym: AQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-0948; 5R21MH107266-02 (NIH)
Record Dates: First submitted 2017-03-13; First posted 2017-03-27 (Actual); Results first posted 2018-06-08 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2017-03

CONDITIONS: Hiv; HIV/AIDS
Keywords: technology; app; YMSM; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: In order to assess the feasibility and acceptability of the app. 20 participants will be enrolled in a one month pilot trial. After being screened for eligibility, the research assistant (RA) will meet with participants in person to explain the study in detail, facilitate app download and login onto participants' phones, and provide an app site tour to highlight features. Participants will complete a baseline demographic and risk assessment administered via a computer assisted survey instrument (CASI). At the end of the one-month field trial, participants will undergo a debriefing session to evaluate their experience using the app, overall satisfaction and any problems they encountered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AllyQuest Pilot (Experimental): The research assistant (RA) will meet with participants in person to explain the study in detail, facilitate app download and login onto participants' phones, and provide an app site tour to highlight features. Participants will complete a baseline demographic and risk assessment administered via a computer assisted survey instrument (CASI). At the end of the one-month field trial, participants will undergo a debriefing session to evaluate their experience using the app, overall satisfaction and any problems they encountered.
  Interventions: Behavioral: AllyQuest

INTERVENTIONS:
Behavioral: AllyQuest — AllyQuest is a novel, high impact secondary prevention intervention delivered via mobile phones to improve linkage and engagement in care among newly diagnosed HIV+ YMSM. The development of this intervention is both timely and vital given the urgency of the ongoing HIV epidemic among YMSM. The features of the intervention aim to target previously identified barriers to care among newly diagnosed youth, namely, low HIV health literacy, lack of social support, and internalized stigma related to their diagnosis.

SUMMARY:
AllyQuest is a novel, high impact secondary prevention intervention delivered via mobile phones to improve linkage and engagement in care among newly diagnosed HIV+ young men who have sex with men (YMSM). The features of the intervention aim to target previously identified barriers to care among newly diagnosed youth, namely, low HIV health literacy, lack of social support, and internalized stigma related to their diagnosis. AllyQuest will be an interactive mobile phone intervention for HIV+ YMSM that utilizes social networking, game-based mechanics and a story-based framework to guide behavior change. Grounded in Social Cognitive Theory, narrative communication and the principles of persuasive technology, the intervention is designed to capitalize on social involvement as a means through which HIV+ YMSM can receive information and social support, experience social norms and reflective appraisals, and feel a sense of connectedness to peers.

DETAILED DESCRIPTION:
Specific Aim 1 Design and develop AllyQuest a novel theory-based mobile health (mHealth) intervention for newly diagnosed HIV+ YMSM. Using an iterative research design the investigators will work with our YABs and Ayogo, a global leader in the application of game psychology and health behavior change, to develop and tailor the intervention content for maximal relevance and usability for newly diagnosed HIV+ YMSM. The investigators will use content within existing evidence based interventions(EBIs) developed for persons living with HIV, including MSM and youth to develop the informational content to be delivered in AllyQuest. Activities from the EBIs will be translated into the daily activities that participants within AllyQuest receive. To maximize intervention appeal and appropriateness for our target population, the investigators will convene two youth advisory boards (YABs) to provide insight and feedback during the intervention development process. The investigators will recruit 4-5 HIV+ YMSM from each site (Chicago and North Carolina) to serve as YAB members over the first year of the study. The investigators will ensure that YAB members are representative of the target population in terms of age, race/ethnicity, sexual orientation/identity, and length of time since diagnosis. At monthly in-person meetings, our two Youth Advisory Boards (YAB) - each consisting of 4 to 5 HIV+ MSM-will evaluate intervention content as it is developed (including imagery and messaging) for acceptability and relevance. Specifically, the investigators will ask YAB members to react to the written tailored content in terms of the content's readability, comprehension, and relevance. The investigators will also elicit the YABs' views on the following areas of intervention design: (a) intervention structure and format [e.g., organization of the intervention, appropriateness and appeal of language/images, ease of navigating the web-based content]; (b) intervention content [e.g., relevance/applicability of intervention content to the population, comprehension of content, interest in the content]; (c) intervention activities [e.g., comprehension of activity instructions, acceptability/relevance of activities, desire to engage in activities]; and (d) overall impressions of the intervention [e.g., overall utility, overall interest, overall enjoyment]. Two YABs are being utilized to ensure maximal diversity of viewpoints and developmental stages during intervention development. During the first six months of year one, YAB members will meet with the research team monthly, as this will be a critical time to develop intervention materials. In addition, web-based meetings and email communication will be used to review materials in between in-person sessions.

Intervention Development and Usability Testing Prototype ideas will be developed in an iterative fashion with Ayogo to develop low-fidelity clickable prototypes that demonstrate the information architecture and high-level features of the application. Members of the research and app development team will conduct internal usability "beta testing" to ensure functionality. After any discovered problems are fixed, 4-5 members of the target population recruited as described above from the North Carolina site and 4-5 members of the target population from the Chicago site will participate in usability testing. Usability testing will assess users comprehension of the educational content, understanding and use of intervention features, and overall impressions of app relevance and appeal. Testing will be conducted in accordance with NIH usability guidelines. Each participant will be asked to meet with a research team member and a member of the development team for a guided, interactive tour through the app. Participants will be asked to share their thoughts and impressions aloud as they move through the different components and features of the app. Audiotapes of the testing sessions along with video tapes of the app screen and participants' hands will be analyzed for patterns of use or usability problems, and results will be compiled into a report for the developers and research team, including any recommendations to address problems identified. Ongoing adjustments require an agile, iterative approach throughout usability testing with members of the target population.

Specific Aim 2 Conduct a one-month pilot trial of AllyQuest with 20 newly diagnosed HIV+ YMSM. To ensure that the features, platform and content of AllyQuest are acceptable to the target population and that there are no technical challenges or user concerns, the investigators will conduct a one-month pilot trial of use. The research assistant (RA) will meet with participants in person to explain the study in detail, facilitate app download and login onto participants' phones, and provide an app site tour to highlight features. Participants will complete a baseline demographic and risk assessment administered via a computer assisted survey instrument (CASI). At the end of the one-month field trial, participants will undergo a debriefing session to evaluate their experience using the app, overall satisfaction and any problems they encountered. Individuals will be instructed to contact the research coordinator immediately to report difficulties with any app components or to report any problems with their phone or phone service. A help link will be embedded within the app that directly links to study staff if assistance is needed. Strategies used in prior team research studies such as employing research staff with training in cultural sensitivity and experience working with HIV+YMSM, providing appropriate monetary incentives for participation in study evaluations, and using available resources to maintain contact will be employed. The investigators will evaluate participant experience with AllyQuest to understand their technology utilization with a specific focus on usability and mechanisms of action that might underlie the potential effectiveness of the intervention (quality/timing of messages, privacy concerns) and quality of the patient-technology relationship (trust, communication, intrusiveness, health promotion). The investigators will also examine barriers and facilitators for implementation. At the end of the one-month pilot trial, participants will complete a quantitative survey administered via a computer assisted survey instrument (CASI). Qualitative exit interviews will allow for a more in-depth and nuanced understanding of intervention acceptability. Interviews will be semistructured and focus on how participants used AllyQuest over the one-month pilot trial and how they perceive that use of the intervention could translate into behavior change.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Diagnosed in the last 12 months
* Assigned male at birth and self identify as male
* Have had sex with another man in the last twelve months
* Own a smart phone
* Between the ages of 16-24

Exclusion Criteria:

* Assigned female at birth
* Non-English speaker
* HIV negative

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — assigned male at birth and self identify as male.
Enrollment: 20 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hightow-Weidman, MD, MPH, Principal Investigator — UNC-CH

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from October, 2016-November, 2016. Participants were recruited from the Cook County Health and Hospitals Systems Infectious Disease Clinic.
Pre-assignment Details: 21 individuals were contacted to recruit them into the study. 20 participants were consented and enrolled, but 21 individuals were assessed for one of the feasibility measures.
Groups:
- AllyQuest Pilot: The research assistant (RA) will meet with participants in person to explain the study in detail, facilitate app download and login onto participants' phones, and provide an app site tour to highlight features. Participants will complete a baseline demographic and risk assessment administered via a computer assisted survey instrument (CASI). At the end of the one-month field trial, participants will undergo a debriefing session to evaluate their experience using the app, overall satisfaction and any problems they encountered.
  AllyQuest is a novel, high impact secondary prevention intervention delivered via mobile phones to improve linkage and engagement in care among newly diagnosed HIV+ YMSM. The features of the intervention aim to target previously identified barriers to care among newly diagnosed youth, namely, low HIV health literacy, lack of social support, and internalized stigma related to their diagnosis.
Period: Overall Study
Arm/Group | AllyQuest Pilot
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AllyQuest Pilot
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Were Enrolled of Those Screened
Description: Feasibility of AllyQuest will be based on recruitment success as measured by the total number of individuals who are screened vs. the total number of individuals who are recruited and subsequently enrolled.
Time Frame: 4 weeks
Population: 21 individuals were assessed for this outcome measure. The number analyzed were those that were recruited and screened for the study, but not enrolled.
Measure: Count of Participants; unit: Participants
Groups:
- AllyQuest Pilot: The research assistant (RA) will meet with participants in person to explain the study in detail, facilitate app download and login onto participants' phones, and provide an app site tour to highlight features. Participants will complete a baseline demographic and risk assessment administered via a computer assisted survey instrument (CASI). At the end of the one-month field trial, participants will undergo a debriefing session to evaluate their experience using the app, overall satisfaction and any problems they encountered.
  AllyQuest: AllyQuest is a novel, high impact secondary prevention intervention delivered via mobile phones to improve linkage and engagement in care among newly diagnosed HIV+ YMSM. The features of the intervention aim to target previously identified barriers to care among newly diagnosed youth, namely, low HIV health literacy, lack of social support, and internalized stigma related to their diagnosis.
Arm/Group | AllyQuest Pilot
Number analyzed (Participants) | 21
Participants | 20

2. Primary Outcome: Number of Participants That Missed Follow up Interviews
Description: Feasibility of AllyQuest will be based retention as measured by the number of missed follow up interviews. Follow up attempts will be documented.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AllyQuest Pilot
Number analyzed (Participants) | 20
Participants | 17

3. Primary Outcome: Average Number of Days Participants Logged in.
Description: Feasibility of AllyQuest will be based on usage as measured by the average number days participants access the app.
Time Frame: 4 weeks
Population: Missing data on 3 participants, hence only reporting data on 17 participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AllyQuest Pilot
Number analyzed (Participants) | 17
days | 21.2 (14.1)

4. Primary Outcome: Number of Individuals Who Enroll But do Not Participate
Description: Feasibility of AllyQuest will be based on the number of individuals who enroll and do not participate.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AllyQuest Pilot
Number analyzed (Participants) | 20
Participants | 3

5. Primary Outcome: Average Total Time in Minutes Participants Spent Using App.
Description: Feasibility of AllyQuest will be based on usage as measured by the average time spent using app.
Time Frame: 4 weeks
Population: Missing data on 3 participants, hence only reporting data on 17 participants.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | AllyQuest Pilot
Number analyzed (Participants) | 17
Minutes | 158.4 (114.1)

6. Primary Outcome: Average Number of App Actions by Participants
Description: Feasibility of AllyQuest will be based on usage as measured by the average number of activities completed (daily quests), articles read, and social posts made.
Time Frame: 4 weeks
Population: Missing data on 3 participants, hence only reporting data on 17 participants.
Measure: Mean (Standard Deviation); unit: Activities completed
Arm/Group | AllyQuest Pilot
Number analyzed (Participants) | 17
Activities completed
  Articles read | 8.8 (7.3)
  Social wall posts | 12.9 (12.5)
  Daily Quests | 15.8 (13.5)

7. Primary Outcome: Average Days Participants Logged Medications.
Description: Feasibility of AllyQuest will be based on usage as measured by the average number of days participants logged their medications in the app.
Time Frame: 4 weeks
Population: Missing data on 3 participants, hence only reporting data on 17 participants.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AllyQuest Pilot
Number analyzed (Participants) | 17
Days | 19.4 (13.2)

8. Secondary Outcome: System Usability Scale Scores
Description: Acceptability of AllyQuest will be measured by the System Usability Scale (SUS). An 11-item, 7-point Likert scale of subjective assessments of usability (1=strongly agree; 7=strongly disagree). The SUS is technology independent and provides a global measure of system satisfaction and sub-scales of usability and learnability.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AllyQuest Pilot
Number analyzed (Participants) | 20
Scores on a scale
  Would use this app frequently | 4.41 (1.18)
  App was easy to use | 4.76 (0.56)
  Felt very confident using the app | 4.47 (1.01)
  App is accurate | 4.53 (1.01)
  App is dependable | 4.53 (0.62)
  Interaction with app is consistent | 4.18 (0.95)
  Found app unnecessarily complex | 1.65 (0.86)
  Would need technical assistance to use app | 1.71 (1.16)
  App features are well integrated | 4.53 (0.80)
  Most people could learn to use app quickly | 4.65 (0.61)
  Found app cumbersome to use | 2.76 (1.64)

9. Secondary Outcome: Client Satisfaction Questionnaire Score
Description: Acceptability of AllyQuest will be assessed using the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 was used to assess global intervention satisfaction. The CSQ-8 has eight items (quality of app, kind of service received from app, app met needs, recommend app to a friend, amount of help received from app, effectiveness of app for dealing with health problem, overall satisfaction, and willingness to use the app again). These domains are assessed on a 4-point response scale with individually specified anchors. Participant responses are scored from 1 to 4, and thus the possible total scores range from 8 to 32. Higher scores indicate greater satisfaction. The CSQ-8 has demonstrated high internal consistency across a large number of studies and has been used to evaluate technology-based interventions
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AllyQuest Pilot
Number analyzed (Participants) | 20
Scores on a scale | 27.8 (5.9)

ADVERSE EVENTS:
Arm/Group | AllyQuest Pilot
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No